CLINICAL TRIAL: NCT01771588
Title: Evaluation of Growth of Pre-Term Infants Fed a Human Milk Fortifier
Brief Title: Human Milk Fortifier - Growth Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08.08.INF
Record Dates: First submitted 2013-01-08; First posted 2013-01-18 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- New human milk fortifier (Experimental): New human milk fortifier
  Interventions: Dietary Supplement: Human milk fortifier
- Currently marketed fortifier (Active Comparator): Currently marketed fortifier
  Interventions: Dietary Supplement: Human milk fortifier
- New human milk fortifier with new Ca source (Experimental): a subgroup of patients will receive the new milk fortifier containing a new source of calcium.
  Interventions: Dietary Supplement: Human milk fortifier

INTERVENTIONS:
Dietary Supplement: Human milk fortifier

SUMMARY:
It it is hypothesized that the growth of preterm infants receiving a new human milk fortifier will be equal or superior to the growth of preterm infants receiving a currently marketed human milk fortifier with a lower protein content.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight ≤1500 g AND/OR gestational age ≤32 weeks (determined by maternal dates, fetal ultrasound, Dubowitz/Ballard examination or a combination thereof)
* Male or female
* Tolerating an enteral intake of human milk, donor milk or a combination at ≥100 mL/kg/d for ≥ 24 h
* Subject is anticipated to receive human milk, donor milk or a combination for ≥ 3 consecutive weeks after having achieved full fortification with volume intake contained between 150 and 180 mL/kg/d.
* Written informed consent has been obtained from the legal representative(s).

Exclusion Criteria:

* Infants with current systemic disease
* Infants with a history of systemic disease
* Any congenital anomalies of the GI tract that significantly interfere with nutrition and growth or previous GI surgery.
* Small size for gestational age (SGA) - body weight ≦ 5th percentile for that gestational age.
* Infants diagnosed with any inherent metabolic disease.
* Infants diagnosed with any chromosomic disease.
* Receiving any commercial formula supplementation to breast milk.
* Receiving steroids at the time of enrollment.
* Participation in another nutritional clinical trial that may affect outcomes of this study.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2011-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Weight gain (g/d) between full strength fortification with full volume intake (day 1) through 21 days of study after that day. | 21 days

CONTACTS AND LOCATIONS:
Locations (11):
- CHR de la Citadelle, Liège, Belgium
- France (7):
  - Hôpital des Enfants - CHU Pellegrin, Bordeaux
  - CHU Caen, Caen
  - CHU Grenoble, Grenoble
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital de la Conception Marseille, Marseille
  - Maternité Régionale, Nancy
  - Hôpital Clocheville Tours, Tours
- Klinikum Ernest von Bergmann, Potsdam, Germany
- Policlinico Mangiagalli e Regina Elena, Milan, Italy
- Kinderspital, Lucerne, Switzerland

REFERENCES:
- [Derived] Rigo J, Hascoet JM, Billeaud C, Picaud JC, Mosca F, Rubio A, Saliba E, Radke M, Simeoni U, Guillois B, de Halleux V, Jaeger J, Ameye L, Hays NP, Spalinger J. Growth and Nutritional Biomarkers of Preterm Infants Fed a New Powdered Human Milk Fortifier: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2017 Oct;65(4):e83-e93. doi: 10.1097/MPG.0000000000001686. PMID 28727654